CLINICAL TRIAL: NCT05102019
Title: Efficacy of the COronary SInus Reducer in Patients With Refractory Angina II
Acronym: COSIRA-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 022-REDUCLN-002
Record Dates: First submitted 2021-10-08; First posted 2021-11-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Refractory Angina
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Arm 1 (treatment arm):Implantation of the Reducer device (Experimental)
  Interventions: Device: Arm 1: treatment with Shockwave Reducer
- Arm 2 (sham-control arm): Control (no device implantation) (Sham Comparator)
  Interventions: Other: Arm 2 (control): Implantation procedure with no device implanted
- Arm 3 (unblinded, non-randomized): Single Arm Registry (Other)
  Interventions: Device: Arm 3 (unblinded, non-randomized): Single arm registry

INTERVENTIONS:
Device: Arm 1: treatment with Shockwave Reducer — Neovasc reducer is an implantable device being evaluated for the alleviation of refractory angina symptoms
  Arms: Arm 1 (treatment arm):Implantation of the Reducer device
Other: Arm 2 (control): Implantation procedure with no device implanted — No device is implanted
  Arms: Arm 2 (sham-control arm): Control (no device implantation)
Device: Arm 3 (unblinded, non-randomized): Single arm registry — Shockwave Reducer is an implantable device being evaluated for the alleviation of refractory angina symptoms
  Arms: Arm 3 (unblinded, non-randomized): Single Arm Registry

SUMMARY:
To demonstrate the safety and effectiveness of the Shockwave Reducer for treatment of patients with refractory angina pectoris treated with maximally tolerated guideline-directed medical therapy who demonstrate objective evidence of reversible myocardial ischemia in the distribution of the left coronary artery and who are deemed unsuitable for revascularization. A non-randomized single-arm registry will further assess the safety and effectiveness of the Shockwave Reducer in selected subjects with reversible myocardial ischemia in the distribution of the right coronary artery and who are deemed unsuitable for revascularization, subjects without documented obstructive coronary disease and abnormal coronary flow reserve (ANOCA), and subjects who cannot complete an exercise tolerance test due to lower limb amputation (above the ankle) or other physiologic condition with documented chronic mobility or balance issues that require the use of a walking aid.

DETAILED DESCRIPTION:
The COSIRA-II study is a multicenter, randomized (1:1 ratio), double-blinded, sham-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is older than 18 years of age
2. Symptomatic coronary artery disease (CAD) with greater than or equal to 90 days of persistent refractory angina pectoris classified as CCS Grade III or IV despite maximally tolerated guideline directed medical therapy as determined by the local heart team and confirmed by a Central Screening Eligibility Committee Note: subjects may also have exertional dyspnea, but the symptoms that limit activity must be anginal in nature (including chest pain, pressure, heaviness, discomfort, with or without radiation to the neck, jaw, shoulders, arms, or other location) and not dyspnea
3. Must have attempted treatment with the maximally tolerated dose of at least three of the four (preferably all four) approved classes of anti-anginal agents: long-acting nitrates, calcium channel blockers (either a dihydropyridine or a non-dihydropyridine), beta blockers, and ranolazine. The regimen must be stable for at least 30 days prior to enrollment, must remain stable from enrollment to randomization, and there must be no intent to change the medical regimen for at least 12 months after randomization Note: If the dose of a medication was increased or decreased for a temporary period and then returned to the original dose, which will then be continued for at least 12 months after randomization, the subject may be immediately enrolled without needing to otherwise requalify
4. Subject has either no treatment options for revascularization by coronary artery bypass grafting or by percutaneous coronary intervention, or is otherwise unsuitable or high risk for revascularization as determined by the local heart team, and confirmed by a Central Screening Eligibility Committee
5. Evidence of either exercise or pharmacologically induced reversible ischemia severity by stress echo, nuclear study, PET, perfusion MRI, CT perfusion, FFR-CT, FFR, iFR, or other non-hyperemic FDA approved tests (such as diastolic hyperaemia free ratio [DRF] or resting full-cycle ratio [RFR] in the distribution of the left coronary artery (LCA), performed within 12 months prior to enrollment and while the patient is maintained on their stable regimen of maximally tolerated doses of anti-anginal medications Note: If the subject has evidence of ischemia in both the LCA and RCA distributions, the extent of ischemia must be greater in the LCA distribution Note: The qualifying assessment must be performed after any myocardial infarction, CABG, or successful PCI within the prior 12 months. If the anti-anginal medication regimen is permanently changed after the assessment of ischemia, the test must be repeated. For subjects with multiple assessments, the one performed closest to enrollment will serve as the qualifying study
6. Functional limitation due to refractory angina as defined by a modified Bruce exercise tolerance test duration of greater than or equal to 2 minutes but less than or equal to 10 minutes, performed while the subject is maintained on their stable regimen of maximally tolerated doses of anti-anginal medications Note: The ETT variability must be less than 20% between last two ETTs performed.
7. Left ventricular ejection fraction (LVEF) greater than or equal to 30% within the 12-months prior to enrollment Note: The LVEF must be reassessed after any intervening myocardial infarction. For subjects with multiple assessments, the most recent LVEF assessment is used as the qualifying test.
8. Subject is willing and able to sign informed consent
9. Subject is willing to comply with the specified follow-up evaluations

Angiographic Inclusion Criteria:

1) Three-vessel coronary angiography performed within 12 months prior to enrollment demonstrating obstructive CAD (visually estimated diameter stenosis of ≥70% or ≥50% - <70% with fractional flow reserve (FFR) value of ≤0.80 or an iFR or other FDA-approved/cleared non-hyperemic physiological assessment (such as DFR or RFR) of ≤0.89 in one or more lesions) in the left coronary artery (main epicardial vessels or branches) that is not suitable for and will not be treated with PCI or CABG as determined by the local heart team Note: The qualifying 3-vessel angiogram must be performed after any myocardial infarction, PCI, or CABG within the 12 months prior to enrollment. For patients with multiple 3-vessel angiograms, the one performed closest to enrollment will serve as the qualifying study

Exclusion Criteria:

1. Recent (within 30 days prior to enrollment) troponin or CKMB positive acute coronary syndrome (NSTEMI or STEMI) Note: subjects with an elevated troponin or CKMB without acute coronary syndrome may still be enrolled
2. Recent successful revascularization by either CABG or PCI within six months prior to enrollment

   Note: Successful revascularization is defined as any CABG procedure, or any PCI procedure with a reduction of one or more lesions to <50% diameter stenosis

   Note: Subjects with successful revascularization by either CABG or PCI that occurred less than six months prior to enrollment may still be approved for participation in the trial if revascularization was completed six months prior to procedure and CSEC approves subject participation
3. Recent unsuccessful PCI (e.g., failed attempt to open a chronic total occlusion) within 30 days prior to enrollment

   Note: Subjects with unsuccessful PCI that occurred less than 30 days prior to enrollment may still be approved for participation in the trial if PCI was completed 30 days prior to procedure and CSEC approves subject participation
4. The predominant manifestation of angina is dyspnea

   Note: some dyspnea may be present with exertion, but the predominant symptom that limits activity must be angina (i.e., chest pain, pressure, tightness, heaviness, or discomfort, with or without radiation to the neck, jaw, shoulders, arms, or other location)
5. Has extra-coronary contributory causes of angina - e.g., untreated hyperthyroidism, untreated anemia (hgb <10 g/dL), uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg despite medications), atrial fibrillation with rapid ventricular response (consistently >100 bpm despite medications) or other tachyarrhythmia, severe aortic stenosis, hypertrophic cardiomyopathy with left ventricular outflow tract obstruction or asymmetric septal hypertrophy (concentric left ventricular hypertrophy is not an exclusion criterion), or epicardial vasospasm disease/coronary artery vasospasm (CAS)/vasospastic angina (VSA)
6. NYHA Class III or IV heart failure (HF), decompensated HF or hospitalization due to HF during the 90 days prior to enrollment
7. Life threatening rhythm disorders or any rhythm disorders that would require future placement of an internal defibrillator and/or pacemaker
8. Severe chronic obstructive pulmonary disease (COPD) as indicated by a forced expiratory volume in one second (FEV1) that is less than 55% of the predicted value, or need for home daytime oxygen or oral steroids
9. Severe valvular heart disease (any valve)
10. Moderate or severe RV dysfunction by echocardiography
11. Pacemaker electrode/lead is present in the coronary sinus
12. A Class I indication is present for an implantable defibrillator or cardiac resynchronization therapy according to ACCF/AHA/HRS guidelines
13. Recent implantation of a new pacemaker or defibrillator lead with electrode in the right atrium within 90 days of enrollment
14. Chronic severe renal failure (estimated eGFR less than 30 mL/min/1.73m2 by the MDRD formula) or subjects on chronic dialysis
15. Known allergy to stainless steel or nickel
16. Any clinical condition that might interfere with the trial protocol or the subject's ability to be compliant with the trial protocol (e.g., active alcohol or drug abuse, dementia, magnetic resonances imaging (MRI) planned within 8 weeks of procedure)
17. Currently enrolled in another investigational device or drug trial that has not reached its primary endpoint or that might clinically interfere with the current trial endpoints or procedures
18. Pregnant or planning pregnancy within the next 12 months (women of reproductive potential must have a negative pregnancy test within 7 days of the procedure)
19. Subject is part of a vulnerable population who, in the judgment of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.
20. Inability to tolerate dual antiplatelet therapy for 6 months if not on a chronic oral anticoagulant, or inability to tolerate a P2Y12 inhibitor for at least 6 months if on a chronic oral anticoagulant
21. Comorbidities limiting life expectancy to less than one year
22. Subject is currently hospitalized for definite or suspected COVID-19
23. Subject has previously been symptomatic with or hospitalized for COVID-19 and has been asymptomatic for <8 weeks prior to enrollment or has not returned to his or her prior baseline (pre-COVID-19) clinical condition
24. Subject is asymptomatic but has had a positive PCR or antigen test for COVID-19 within the past 4 weeks prior to enrollment

Angiographic/Hemodynamic Exclusion Criteria:

1) Coronary anatomy amenable to revascularization of ischemic myocardial territory by either PCI or CABG with at least moderate likelihood of long-term alleviation of angina or angina equivalent symptoms, as per the assessment of the local heart team.

Note: If a pathway to coronary revascularization is present which, in the opinion of the local heart team, is reasonably low risk and reasonably likely to provide long-term symptom relief and the subject refuses the revascularization procedure, the patient is ineligible for randomization

Procedural Angiographic/Hemodynamic Randomization Exclusion Criteria:

1. Mean right atrial pressure greater than 15 mmHg assessed during the final screening procedure for eligibility assessment and potential randomization
2. Anomalous or abnormal CS anatomy (e.g., tortuosity, aberrant branch, persistent left superior vena cava [SVC]) as demonstrated by angiogram
3. The CS diameter at the most proximal end of the planned implant region (2-4 cm distal to the coronary sinus ostium) is less than 9.5 mm or greater than 13.0 mm

Single-arm Registry (Unblinded, Non-Randomized Treatment Arm) Inclusion/Exclusion Criteria:

Subject can be included in the single-arm registry if they fall into one of the three categories with inclusions and exclusion criteria as described below.

Predominant right coronary disease subjects (RCA):

1. Reversible ischemia: Subjects with evidence of either exercise or pharmacologically induced reversible ischemia by stress echo, nuclear study, PET, perfusion MRI, CT perfusion, FFR-CT, FFR, iFR, or other non-hyperemic FDA approved or cleared tests (such as DFR or RFR) in the distribution of the right coronary artery (RCA), performed within 12 months prior to enrollment.

   Note: If the subject has evidence of ischemia in both the LCA and RCA distributions, the extent of ischemia must be greater in the RCA distribution

   Note: The qualifying assessment must be performed after any myocardial infarction, CABG, or successful PCI within the prior 12 months. If the anti-anginal medication regimen is permanently changed after the assessment of ischemia, the test must be repeated. For subjects with multiple assessments, the one performed closest to enrollment will serve as the qualifying study
2. Obstructive CAD: Three-vessel coronary angiography performed within the 12 months prior to enrollment demonstrating obstructive CAD (visually assessed diameter stenosis of ≥70% or ≥50% - <70% with fractional flow reserve (FFR) value of ≤0.80 or an iFR or other FDA-approved/cleared non-hyperemic physiological assessment (such as DFR or RFR) of ≤0.89 in one or more lesions) in the RCA (main epicardial vessels or branches) that is not suitable for and will not be treated with PCI or CABG as determined by the local heart team.

   Note: The qualifying assessment must be performed after any myocardial infarction, PCI or CABG within the prior 12 months. For subjects with multiple assessments, the one performed closest to enrollment will serve as the qualifying study
3. In addition to the above inclusion criteria, subjects must meet all inclusion criteria (except clinical inclusion #5 and angiographic inclusion #1) and none of the exclusion criteria of the main randomized trial

Non-obstructive coronary artery disease subjects (ANOCA)

1. Abnormal Coronary Flow Reserve (CFR): subjects must have either abnormal PET CFR (< 2.0) or abnormal invasive CFR (<2.5) in at least one main epicardial coronary artery performed within 12 months prior to enrollment

   Note: Subjects may or may not have evidence of either exercise or pharmacologically induced reversible ischemia by stress echo, nuclear study, PET, perfusion MRI, or CT perfusion
2. Non-obstructive CAD: subjects have non-obstructive coronary disease (estimated diameter stenosis in all coronary lesions is <50% and (if performed) FFR ≥0.81 or a non-hyperemic test is ≥0.90) demonstrated on three-vessel coronary angiography performed within the 12 months prior to enrollment. If an estimated diameter stenosis is ≥50% to <70%, the patient may still qualify if FFR ≥0.81 or a non-hyperemic test is ≥0.90 in that vessel. If both FFR and a non-hyperemic test are performed, both must be negative.

   Note: The qualifying 3-vessel angiogram must be performed after any myocardial infarction, PCI or CABG within the 12 months prior to enrollment. For patients with multiple 3-vessel angiograms, the one performed closest to enrollment will serve as the qualifying study
3. In addition to the above inclusion criteria, subjects must meet all inclusion criteria (except clinical inclusion #5 and angiographic inclusion #1) and none of the exclusion criteria of the main randomized trial

Subjects unable to complete ETT

1. Subjects must be unable to complete the required COSIRA-II exercise tolerance test due to lower limb amputation (above the ankle) or other physiologic condition with documented chronic mobility or balance issues that require the use of a walking aid (e.g., wheelchair, cane, rollator, crutches, or knee walker).
2. In addition to the above inclusion criteria, subjects must meet all inclusion criteria (except clinical inclusion #6) and none of the exclusion criteria of the main randomized trial

Prior to inclusion in single-arm registry, all subjects will be reviewed by the Central Screening Eligibility Committee to ensure that they meet registry inclusion criteria and are not eligible for enrollment into the randomized study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 6 months
  Change in total exercise duration in a modified Bruce treadmill exercise tolerance testing evaluation in the Treatment arm compared to Sham-control arm.
Safety Events | 6 months
  The rate of occurrence of a composite of death, myocardial infarction (MI), pericardial effusion requiring surgical or percutaneous intervention, device embolization, or BARC 3 or 5 bleeding evaluation in the Treatment arm compared to the Sham-control arm.

SECONDARY OUTCOMES:
Canadian Cardiovascular Society (CCS) Angina Score | 6 months
  Improvement by greater than or equal to 1 CCS angina grade. The CCS grading system for angina is a clinical tool used by doctors to assess the degree of severity of a patient's angina. Possible scores range from Class 0 (asymptomatic angina) to Class IV (angina at rest).
Canadian Cardiovascular Society (CCS) Angina Score | 6 months
  Improvement by greater than or equal to 2 CCS angina grades. The CCS grading system for angina is a clinical tool used by doctors to assess the degree of severity of a patient's angina. Possible scores range from Class 0 (asymptomatic angina) to Class IV (angina at rest).
Seattle Angina Questionnaire (SAQ) Score | 6 months
  Change in Angina Stability domain score from the Seattle Angina Questionnaire (SAQ). The Seattle Angina Questionnaire (SAQ) is a disease-specific questionnaire used to quantify patients' symptoms of angina and the extent to which their angina affects their functioning and quality of life. Possible scores range from 0 (daily angina) to 100 (no angina). Lower scores indicate worse angina symptoms.

OTHER OUTCOMES:
Canadian Cardiovascular Society (CCS) Angina Score | 12 months, 2 years, 3 years, 4 years, and 5 years
  Improvement by greater than or equal to 1 and greater than or equal to 2 CCS angina grades compared to baseline. The CCS grading system for angina is a clinical tool used by doctors to assess the degree of severity of a patient's angina. Possible scores range from Class 0 (asymptomatic angina) to Class IV (angina at rest).
Angina Burden | 6 and 12 months
  Angina frequency and burden compared to baseline
Activity | 6 and 12 months
  Measure of activity assessed by actigraphy compared to baseline
Exercise Tolerance Testing | 6 and 12 months
  Change in ETT parameters compared to baseline
Exercise Tolerance Testing | 12 months
  Change in total exercise duration compared to baseline
Doctor Visits | 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Number of unplanned office visits due for angina, and any hospitalizations or emergency department visits (for angina, non-angina cardiovascular causes) post procedure compared to baseline
Exercise Tolerance Testing | 6 and 12 months
  Total exercise duration
Seattle Angina Questionnaire (SAQ) Score | 6 month, 12 month, 2 years, 3 years, 4 years, and 5 years
  Change in other Seattle Angina Questionnaire (SAQ) domain scores compared to baseline. The Seattle Angina Questionnaire (SAQ) is a disease-specific questionnaire used to quantify patients' symptoms of angina and the extent to which their angina affects their functioning and quality of life. Possible scores range from 0 (daily angina) to 100 (no angina). Lower scores indicate worse angina symptoms.
Adverse Events | 30 day, 6 month, 12 month, 2 years, 3 years, 4 years, and 5 years
  Number of deaths, myocardial infarctions, strokes, unplanned revascularization procedures in-hospital, at 30 days, 3 months, 6 months, 12 months and annually post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Henry, MD, Principal Investigator — The Christ Hospital Health Network; Gregg W Stone, MD, Principal Investigator — Mt. Sinai Heart Health
Locations (91):
- United States (69):
  - Mayo Clinic, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - Long Beach VA Medical Center, Long Beach, California
  - Cedars-Sinai, Los Angeles, California
  - UCSD, San Diego, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - UCSF, San Francisco, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - South Denver Cardiology Associates, Littleton, Colorado
  - Yale University, New Haven, Connecticut
  - MedStar Cardiovascular Research Network, Washington D.C., District of Columbia
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Mount Sinai Miami, Miami Beach, Florida
  - NCH Healthcare - Naples, Naples, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Tampa General - USF Cardiology, Tampa, Florida
  - Emory Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia, Gainesville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Ascension St. Vincent Heart Center, Carmel, Indiana
  - Community Hospital - Munster, Munster, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford St. Johns, Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Henry Ford Providence, Southfield, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Saint Luke's Hospital, Kansas City, Missouri
  - Hackensack University, Hackensack, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - NYU Langone, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Novant Health, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Ascension St. John, Tulsa, Oklahoma
  - Providence Heart Institute, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt Heart, Nashville, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
  - Medical City Fort Worth, Fort Worth, Texas
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - Houston Methodist, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Hospital of San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Advocate Aurora Research Institute, Milwaukee, Wisconsin
- Canada (5):
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital (UHN), Toronto, Ontario
  - CHUM, Montreal, Quebec
  - IUCPQ-Ulaval, Québec, Quebec
- United Kingdom (17):
  - Essex Cardiothoracic Centre, Basildon
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Bristol Heart Institute, Bristol
  - Dorset County Hospital NHS Foundation Trust, Dorchester
  - Kettering General Hospital, Kettering
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Barts Health Centre, London
  - Royal Free Hospital, London
  - St. Thomas Hospital, London
  - King's College Hospital, London
  - Royal Brompton Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospital, Nottingham
  - Oxford University Hospital, Oxford
  - Royal Bournemouth Hospital, Poole
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verheye S, Jolicoeur EM, Behan MW, Pettersson T, Sainsbury P, Hill J, Vrolix M, Agostoni P, Engstrom T, Labinaz M, de Silva R, Schwartz M, Meyten N, Uren NG, Doucet S, Tanguay JF, Lindsay S, Henry TD, White CJ, Edelman ER, Banai S. Efficacy of a device to narrow the coronary sinus in refractory angina. N Engl J Med. 2015 Feb 5;372(6):519-27. doi: 10.1056/NEJMoa1402556. PMID 25651246
- [Derived] Bober RM, Johnson NP. How might coronary sinus reducer treatment change myocardial perfusion? J Nucl Cardiol. 2024 Mar;33:101828. doi: 10.1016/j.nuclcard.2024.101828. Epub 2024 Feb 21. No abstract available. PMID 38395338